CLINICAL TRIAL: NCT01638455
Title: Noninvasive Parameter Testing With Pulse CO-Oximetry and Measurement of Blood Constituents With In-Vitro Analyzers
Brief Title: Pulse CO-Oximetry Noninvasive Monitoring and Laboratory Measurements of Subject Blood Samples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: Masimo-Noninvasive 1
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Various Comorbidities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Test Group (Experimental): All subjects will be enrolled in the test group and will receive the noninvasive device
  Interventions: Device: Noninvasive device

INTERVENTIONS:
Device: Noninvasive device — Noninvasive device

SUMMARY:
Characterize Masimo noninvasive technology in spot check reading on subjects and make comparison to invasive blood sampling tested on reference analyzers.

DETAILED DESCRIPTION:
Noninvasive readings from subjects done according to manufacturer's directions of use compared to simultaneously derived blood samples measured on in vitro analyzers

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any age ≥ 3 kg.
* Subjects may include healthy volunteers, outpatient or inpatient populations

Exclusion Criteria:

* Subjects with skin abnormalities at the planned application sites that may interfere with sensor application or trans-illumination of the site, such as burns, scar tissue, nail polish, acrylic nails, infections, etc.
* Subjects deemed not suitable for study at the discretion of the investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2776 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2016-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo, Irvine, California, United States